CLINICAL TRIAL: NCT01124331
Title: Appropriate Levels of Oxygen Saturation for Extremely Preterm Infants: Prospective Individual Patient Data Meta-analysis
Brief Title: Appropriate Oxygen Levels for Extremely Preterm Infants: a Prospective Meta-analysis
Acronym: NeOProM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: University of Otago (Other); University of Oxford (Other); University of Pennsylvania (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NeOProM
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Infant, Premature, Diseases; Bronchopulmonary Dysplasia; Retinopathy of Prematurity; Infant, Newborn, Diseases; Infant, Very Low Birth Weight
Keywords: prospective meta-analysis; preterm infant; pulse oximetry; oxygen saturation
MeSH Terms: conditions — Infant, Premature, Diseases; Bronchopulmonary Dysplasia; Retinopathy of Prematurity; Infant, Newborn, Diseases; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Oxygen saturation (Experimental): Higher (SpO2 91-95%) functional oxygen saturation target range from birth, or soon thereafter, for durations as specified in each trial protocol.
  Interventions: Procedure: Higher oxygen saturation target range (91%-95%)
- Lower oxygen saturation (Active Comparator): Lower (SpO2 85-89%) functional oxygen saturation target range from birth, or soon thereafter, for durations as specified in each trial protocol.
  Interventions: Procedure: Lower oxygen saturation (85%-89%)

INTERVENTIONS:
Procedure: Higher oxygen saturation target range (91%-95%) — higher (SpO2 91-95%) functional oxygen saturation target range from birth, or soon thereafter
  Arms: High Oxygen saturation
Procedure: Lower oxygen saturation (85%-89%) — Lower (SpO2 85%-89%)functional oxygen saturation target range from birth, or soon thereafter
  Arms: Lower oxygen saturation

SUMMARY:
The primary question to be addressed by this study is: compared with a functional oxygen saturation level (SpO2) of 91-95%, does targeting SpO2 85-89% in extremely preterm infants from birth or soon after, result in a difference in mortality or major disability in survivors by 2 years corrected age (defined as gestational age plus chronological age)?

DETAILED DESCRIPTION:
Oxygen has been used in the care of small and sick newborn babies for over 60 years. However, to date there has been no reliable evidence to guide clinicians regarding what is the best level to target oxygen saturation in preterm infants to balance the four competing risks of mortality, lung disease, eye damage and developmental disability.

Five high quality randomised controlled trials are now underway assessing two different levels of oxygen saturation targeting (USA - SUPPORT; Australia - BOOST II; New Zealand - BOOST NZ; UK - BOOST II UK; Canada - COT). The value of these gold-standard trials can be further enhanced when, with careful planning, they are synthesised into a prospective meta-analysis (PMA). A PMA is one where trials are identified for inclusion in the analysis before any of the individual results are known.

We have established the Neonatal Oxygenation Prospective Meta-analysis (NeOProM) Collaboration, comprising the investigators of these five trials and a methodology team. The trials are sufficiently similar with respect to design, participants and intervention and, with planning, will have enough common outcome measures to enable their results to be prospectively meta-analysed. Together they have a combined sample size of almost 5000 enrolled infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants < 28wks gestation

Exclusion Criteria:

* Infants > 28wks gestation

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4965 (Actual)
Dates: Start 2005-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
composite outcome of death or major disability by 18-24 months corrected age | by 18-24 months corrected age (gestational age plus chronological age)
  Major disability is defined as any of the following:
  * Bayley-III Developmental Assessment cognitive score <85 and/or language score <85
  * Severe visual loss
  * Cerebral palsy with Gross Motor Function Classification System (GMFCS) level 2 or higher or Manual Ability Classification System (MACS) level 2 or higher at 18-24 months postmenstrual age
  * Deafness requiring hearing aids

SECONDARY OUTCOMES:
Retinopathy of prematurity (ROP) treatment by laser photocoagulation or cryotherapy or anti-VEGF injection | at 18-24 months corrected age
measures of respiratory support | 36 weeks postmenstrual age
  • Measures of respiratory support, including the following separate outcomes a. supplemental oxygen requirement at 36 weeks postmenstrual age, b. postmenstrual age ceased endotracheal intubation, c. postmenstrual age ceased continuous positive airway pressure (CPAP), d. postmenstrual age ceased supplemental oxygen, e. postmenstrual age ceased home oxygen (if received).
Patent ductus arteriosus diagnosed by ultrasound and receiving medical treatment | at 18-24 months corrected age
Patent ductus arteriosus receiving surgical treatment | at 18-24 months corrected age
Weight z-score based on WHO percentile charts (WHO Multicentre Growth Reference Study Group, 2006) | 18-24 months corrected age
Weight z-score based on WHO percentile charts (WHO Multicentre Growth Reference Study Group, 2006) | at 36 weeks' postmenstrual age and discharge home
Re-admissions to hospital | up to 18-24 months postmenstrual age
Cerebral palsy with GMFCS level 2 or higher or MACS level 2 or higher at 18-24 months corrected age | at 18-24 months corrected age
Severe visual impairment (cannot fixate or is legally blind:<6/60 vision , 1.3 logMAR in both eyes or equivalent as defined by trial) | at 18-24 months corrected age
deafness requiring hearing aids | at 18-24 months corrected age
Bayley-III Developmental Assessment cognitive score <85 and/or language score <85 | 2 years corrected age
death | at 18-24 months corrected age

OTHER OUTCOMES:
Subgroup analyses will be undertaken on all pre-specified primary and secondary outcomes. | at 18-24 months corrected age
  Subgroups:
  * Gestational age
    * less than 26 weeks
    * greater than or equal to 26 weeks
  * Inborn or outborn
  * Use of any antenatal corticosteroids = yes if any of the following
    * incomplete, less than 24 hours before birth
    * complete
    * more than 7 days before birth
    * started less than 24h before birth
    * started 24h or more before birth
  * Male or female gender
  * Small for gestation age
    * birth weight below trialist defined cut-point
    * birth weight less than 10th percentile using WHO centile charts
  * Multiple or singleton birth
  * Mode of delivery
    * Vaginal if any of the following: vaginal, vaginal-cephalic, vaginal-breech
    * Caesarean if any of the following: caesarean, caesarean section before onset of labour, caesarean section after onset of labour, caesarean section
  * Time of intervention commencement
    * less than 6 hours after birth
    * 6 hours or more after birth
  * Oximeter calibration software
    * original
    * revised

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Askie, Principal Investigator — National Health and Medical Research Council, Australia
Locations (9):
- Australia (9):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Royal Prince Alfred Hospital Women and Babies, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Royal North Shore Hospital, NSW, St Leonards, New South Wales
  - Westmead Hospital,, Westmead, New South Wales
  - Royal Brisbane Women's Hospital, Brisbane, Queensland
  - Royal Women's Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria

REFERENCES:
- [Background] Askie LM, Brocklehurst P, Darlow BA, Finer N, Schmidt B, Tarnow-Mordi W; NeOProM Collaborative Group. NeOProM: Neonatal Oxygenation Prospective Meta-analysis Collaboration study protocol. BMC Pediatr. 2011 Jan 17;11:6. doi: 10.1186/1471-2431-11-6. PMID 21235822
- [Result] Askie LM, Darlow BA, Finer N, Schmidt B, Stenson B, Tarnow-Mordi W, Davis PG, Carlo WA, Brocklehurst P, Davies LC, Das A, Rich W, Gantz MG, Roberts RS, Whyte RK, Costantini L, Poets C, Asztalos E, Battin M, Halliday HL, Marlow N, Tin W, King A, Juszczak E, Morley CJ, Doyle LW, Gebski V, Hunter KE, Simes RJ; Neonatal Oxygenation Prospective Meta-analysis (NeOProM) Collaboration. Association Between Oxygen Saturation Targeting and Death or Disability in Extremely Preterm Infants in the Neonatal Oxygenation Prospective Meta-analysis Collaboration. JAMA. 2018 Jun 5;319(21):2190-2201. doi: 10.1001/jama.2018.5725. PMID 29872859